CLINICAL TRIAL: NCT05924906
Title: Phase 1a/1b, First-in-Human, Open Label, Dose Escalation and Dose Expansion Study of NB002, a Multifunctional TIM-3 Blocking Antibody, in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Dose Escalation and Expansion Study of NB002 in Participants With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Neologics Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NB002-101
Record Dates: First submitted 2023-05-25; First posted 2023-06-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: BOIN design dose escalation scheme for phase Ia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- NB002 dose level 1 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002
- NB002 dose level 2 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002
- NB002 dose level 3 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002
- NB002 dose level 4 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002
- NB002 dose level 5 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002
- NB002 dose level 6 (Experimental): NB002 is a recombinant humanized IgG1 monoclonal antibody
  Interventions: Drug: NB002

INTERVENTIONS:
Drug: NB002 — Strength: 100 mg:5 mL solution in a single-use vial Administration: intravenous infusion

SUMMARY:
This study is a first-in-human, multicenter, open label, uncontrolled, non-randomized, phase 1a/1b study, to evaluate the safety, tolerability, and preliminary antitumor activity of NB002 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a first-in-human, multicenter, open-label, uncontrolled, non-randomized, phase 1a/1b study. The study consists of a dose escalation part and a dose expansion part. In the escalation part, the primary objectives are to characterize the safety, tolerability, and dose-limiting toxicities (DLTs) to establish a preliminary recommended Phase 2 dose (RP2D) and/or a maximum tolerated dose (MTD) or maximum administered dose (MAD) of NB002. The expansion part is to further evaluate the safety and tolerability of NB002 at the RDE dose established in the dose escalation part and to explore antitumor activity in the selected population. All subjects will be treated with NB002 via IV infusion at predefined dose levels Q3W on Day 1 of each 21-day Cycle.

The design of the dose escalation part will be provided below. Further details on dose expansion part will be updated later once more information on potentially benefiting tumor types is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of signing informed consent.
2. Diagnosis of histological or cytological confirmed locally advanced, recurrent and/or metastatic solid tumors that failed to respond to standard therapy, intolerant/refractory to currently available local therapies, or for whom no appropriate therapies are available (based on the judgement of the Investigator).
3. Measurable or non-measurable disease according to RECIST 1.1 in dose escalation stage and at least one measurable lesion is necessary for dose expansion stage.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1, and anticipated life expectancy of ≥ 3 months.
5. Adequate hematologic function based on the following (with no blood transfusion or hematopoietic stimulating factor therapy within 14 days prior to study drug administration):

   1. ANC≥1.2 ×10^9/L
   2. Platelet count ≥75×10^9/L
   3. Hemoglobin ≥8.0 g/dL
6. Adequate coagulation parameters based on the following:

   1. Prothrombin Time-International Normalized Ratio (PT-INR) ≤1.5×ULN (upper limit of normal), unless coumarin derivatives are used.
   2. Activated partial thromboplastin time (aPTT) ≤1.5×ULN. Subjects on anticoagulants may have coagulation parameters that exceed the criteria defined above.
7. Adequate hepatic function based on the following:

   1. Total bilirubin (TBIL) ≤1.5 × ULN and/or isolated elevations of indirect bilirubin are eligible for study participation.
   2. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤3 × ULN (≤5 × ULN for subjects with known hepatic metastases).
8. Adequate renal function based on serum creatinine clearance ≥30 mL/min (normal to moderate renal impairment) as determined by Cockcroft-Gault equation.
9. A female patient is eligible to participate if she is not pregnant or breastfeeding, and

   * is not a WOCBP or
   * A WOCBP must have a negative pregnancy test within 72 hours before the first dose of study drug administration, and additional pregnancy testing during and after study drug as defined in the SOA .
   * A WOCBP must consent to use highly effective contraceptive methods or abstain from heterosexual activity from screening through 120 days following the last dose of study treatment.
10. Fertile male subjects, defined as all males physiologically capable of conceiving offspring, with their WOCBP partner(s) must agree to use highly effective contraception. Sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to abstain from sexual intercourse or use barrier contraception from Screening through 120 days following the last dose of study treatment.
11. Ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria:

1. Inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first administration of study drug.
2. Has had a known or suspected hypersensitivity reaction to treatment with a mAb and/or the excipients of NB002.
3. Prior treatment with other TIM-3 inhibitors (e.g., mAbs).
4. Prior palliative radiotherapy within 1 week of start of study treatment. Subjects must have recovered (CTCAE Grade ≤1) from all radiation-related toxicities.
5. Any antitumor agent for the primary malignancy without delayed toxicity within 4 weeks or 5 half-lives, whichever is shorter, prior to first administration of study drug, except for Nitrosoureas and mitomycin C within 6 weeks prior to first administration of study drug and during study.
6. Active CNS metastases, however, subjects who have undergone definitive radiation and/or surgery for the treatment of CNS metastases, who are stable by radiographic and clinical (neurological) assessment (performed within 4 weeks prior to first trial drug administration), and who are no longer taking pharmacologic doses of corticosteroids are eligible; subjects with leptomeningeal metastases or primary CNS malignancies (such as glioma, glioblastoma) are not eligible.
7. Evidence of metastatic ileus on computed tomography (CT) scan.
8. Patients with concurrent hematologic malignancies.
9. Known active or prior infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV), or hepatitis C virus (HCV).
10. Any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks prior to first administration of study drug.
11. Patients with an active, known or suspected autoimmune disease, or a documented history of autoimmune disease or syndrome, requiring systemic steroids or other immunosuppressive medications. procedure is allowed if all other inclusion/exclusion criteria are met.
12. History of organ transplantation (e.g., stem cell or solid organ transplant)
13. A significant pulmonary disease or condition.
14. Patients with a current or recent (within 6 months) significant gastrointestinal (GI) disease or condition.
15. History of immune-related toxicity during prior treatment with an immune checkpoint inhibitor (ICI, e.g., PD-1/PD-L1 or CTLA-4 inhibitor), including any grade ≥3, and neurologic and/or ocular immune-related toxicity, pneumonitis, or cardiomyopathy of any grade that necessitated permanent discontinuation of that therapy. Patients with other Grade 1-2 immune-related toxicities on prior ICI therapy that have resolved are NOT excluded. Endocrine immune-related toxicities of grade <3 are allowed, as long as they are controlled and/or asymptomatic. Substitution therapy following an immune-related endocrinopathy is allowed.
16. Unresolved > Grade 1 toxicity associated with any prior antitumor therapy except for persistent Grade 2 alopecia, peripheral neuropathy, decreased hemoglobin, lymphopenia, hypomagnesemia, and/or end-organ failure being adequately managed by hormone replacement therapy:
17. Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to first administration of study drug unless adequately treated and considered by the Investigator to be stable. Active uncontrolled bleeding or a known bleeding diathesis.
18. Vaccination with live vaccine(s) within 1 month prior to administration.
19. Baseline QT interval corrected with Fridericia's method (QTcF) >470 ms (average of triplicate electrocardiograms [ECG]).
20. Unstable or severe uncontrolled medical condition (e.g., uncontrolled diabetes), psychiatric illness/social situations, or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE), serious adverse events (SAE) | Up to 12 months
  AEs will be evaluated by the investigator, according to criteria outlined in the NCI CTCAE version 5.0
Number of participants with dose-limiting toxicity (DLT), as defined in the protoocol | 21 days
  All toxicities will be graded according to NCI CTCAE version 5.0 based on the investigator assessment. The DLT window of observation will be during Cycle 1 (21 days).

SECONDARY OUTCOMES:
Pharmacokinetics of NB002: Maximum plasma concentration of the study drug (Cmax) | Up to 12 months
  Maximum observed plasma or serum concentration.
Pharmacokinetics of NB002: Time to maximum concentration (Tmax) | Up to 12 months
  Time to maximum concentration.
Pharmacokinetics of NB002: Minimum plasma concentration of the study drug (Cmin) | Up to 12 months
  Minimum observed plasma or serum concentration over the dose interval.
Pharmacokinetics of NB002: Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC0-t) | Up to 12 months
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Objective response (OR) | Up to 12 months
  Complete response (CR) or partial response (PR), as defined by RECIST v1.1
Progression free survival (PFS) | Up to 12 months
  The time from first dose of study intervention until the date of objective disease progression or death
Duration of response (DOR) | Up to 12 months
  The time from first response according to RECIST v1.1 until progression or death
Pharmacodynamics (PD) activity (Level of binding of NB002 to TIM-3 ) | Up to approximately 3 months
  Receptor occupancy in peripheral blood mononuclear cells (PBMCs) or whole fresh blood
Immunogenicity of NB002 | Up to 12 months
  The number and percentage of participants who develop detectable anti-drug antibodies (ADA).

IPD SHARING:
Plan to Share IPD: No